CLINICAL TRIAL: NCT04063917
Title: An Initial Investigation of the Safety and Tolerability of Transcutaneous Stimulation of the Hypoglossal Nerve for the Treatment of Primary Snoring and Mild Sleep Apnea Using the ZENS Transcutaneous Nerve Stimulator (PLUTO)
Brief Title: Safety, and Tolerability of the ZENS Device (PLUTO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zennea Technologies Inc. (Industry)
Collaborators: University of Calgary (Other); Interior Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CIP-001
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Snoring; Obstructive Sleep Apnea
Keywords: Sleep Apnea; Snoring
MeSH Terms: conditions — Snoring; Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Multi-center, open label randomized 2x2 cross-over sleep study of the ZENS transcutaneous hypoglossal nerve stimulator in the "ON" (active) versus "OFF" (passive) setting during a single over-night sleep study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence 1 (Experimental): Participants allocated to Sequence 1 will complete the overnight sleep study with the ZENS device "ON" for the first half and "OFF" for the second half.
  Interventions: Device: ZENS
- Sequence 2 (Experimental): Participants allocated to Sequence 1 will complete the overnight sleep study with the ZENS device "OFF" for the first half and "ON" for the second half
  Interventions: Device: ZENS

INTERVENTIONS:
Device: ZENS — ZENS transcutaneous nerve stimulator (ZENS Device), a wearable and non-invasive device which stimulates nerves in the neck to reduce airway obstruction and maintain muscular tension while sleeping to reduce snoring severity.

SUMMARY:
The primary objective of the PLUTO study is to evaluate the safety and tolerability of the ZENS transcutaneous nerve stimulator device in primary snorers and those with mild obstructive sleep apnea. The study will assess the impact of ZENS on snoring frequency, duration, and other relevant sleep parameters. The intended purpose of the investigational device is to deliver a transcutaneous electrical stimulation signal to the hypoglossal nerve in the "ON" phase in order to alter the apnea hypopnea index (AHI), as well as mean snoring burden (intensity, duration), and to deliver no signal in the "OFF" phase of the study as a means for comparison. Subjects utilizing the ZENS Device will experience a reduction in snoring during the "ON" versus "OFF" phase, as quantified by a reduction in the percentage of time per hour of snoring (≥40 dB) in the active ZENS Device ("ON" phase) versus the inactive ZENS Device ("OFF" phase).

DETAILED DESCRIPTION:
After indicating their consent to contact and signing an Informed Consent Form, potential participants will undergo a screening assessment that includes a review of their medical history, a focused physical exam, and a level 3 at-home sleep test (Sagatech SnoreSat Sleep Recorder, Philips Alice OneNight or equivalent), if not already available in the medical records). At the screening visit potential participants' eligibility for the study will be evaluated against the study inclusion and exclusion criteria.

Following confirmation of eligibility, up to 45 (n=45) participants will be scheduled for their overnight in-laboratory PSG, which must occur no more than 12 weeks after screening has taken place. A final determination of eligibility and "enrollment" is completed when inclusion and exclusion criteria are verified on the day of the study visit. Those who do not meet inclusion and exclusion criteria on the day of the study will be deemed "screening failures".

Participants will wear the ZENS Device for the 8 to 12-hour overnight in-laboratory polysomnography assessment. Participants will be monitored for and asked about any adverse events and device effects that they experience during the overnight sleep study.

Participants will be contacted by the site via telephone 24 to 96 hours after the overnight sleep study to determine if any adverse events and device effects were experienced late after the overnight polysomnography. After the telephone follow-up, participation in the study is complete.

ELIGIBILITY:
Inclusion:

1. Adult (age of majority).
2. Willing and able to provide written informed consent.
3. BMI <35.
4. Neck circumference <18 inches.
5. History of disruptive snoring for most of the night, 12 or more of the last 14 nights.
6. Level 3 at-home sleep test (Sagatech SnoreSat Sleep Recorder, Philips Alice OneNight or equivalent) recording from the past 12 months (prior to enrolment) with more than 4 hours of both oximetry and flow data for review; or willing to undergo a level 3 sleep test prior to overnight in-laboratory polysomnography assessment. The respiratory disturbance index (RDI) must be <15events/hour.
7. Ability and willingness to shave significant facial hair (i.e. be clean shaven) for the overnight visit; and to cease wearing cosmetic products and/or moisturizing cream and/or remove excessive oil in the chin / jaw region (i.e. be clean skinned) for the overnight visit; and to wear clothing that covers the chest (e.g. a t-shirt) for the duration of the overnight visit.
8. Willing to participate in overnight portion of study without use of another snoring/OSA treatment (CPAP, oral appliance) in the 72 hours prior to the overnight visit.
9. Willing to refrain from use of alcohol, sedative hypnotics, or recreational drugs for 24 hours prior to and during the study.

Exclusion:

1. Prior diagnosis of moderate or severe OSA (AASM defines OSA severity as: Mild=AHI ≥5 and <15; Moderate=AHI ≥15 and <30; Severe = ≥30/hour).
2. Known sleep disturbance other than snoring (insomnia, parasomnia, narcolepsy, restless legs syndrome, circadian rhythm disorder, or other disorder likely to interfere with the study).
3. Fixed anatomical abnormality of the upper airway (e.g. history of head or neck trauma, head and neck malignancy, previous tracheotomy, subglottic stenosis, deformed uvula, aglossia) from trauma, malignancy, prior surgery, or congenital condition.
4. Individuals with a history of severe nasal obstruction due to anatomical problems such as deviated septum, previously broken nose or non-anatomical factors such as chronic rhinitis or nasal polyposis.
5. Enflamed/enlarged tonsils.
6. Use of another snoring treatment (CPAP, medication or oral appliance) in the 72 hours prior to the overnight visit.
7. Anatomic neck or skin abnormalities likely to interfere with fixation of the ZENS Device.
8. Presence of an implantable medical device susceptible to electrical interference (e.g. pacemaker or defibrillator).
9. History of epilepsy.
10. Use of sedatives, hypnotics, recreational drug or alcohol in the 24 hours prior to the study.
11. Known allergy to medical tape.
12. Any severe skin condition affecting the head and neck likely to be aggravated by adhesives (e.g. psoriasis, eczema).
13. Recent surgery to the face or neck (i.e. within the past 5 years).
14. Inability to wear something on the neck or tolerate PSG procedure.
15. Pregnancy.
16. Any other criteria, which would make the participant unsuitable to participate in this study as determined by the site Principal Investigator (e.g. uncontrolled drug and/or alcohol addiction, extreme frailty, comorbidities, ongoing medication regimen, cognitive ability to follow instructions, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Percent change in loud snoring time | up to 5 hours
  The percentage change in snoring time in the "ON" versus "OFF" period

SECONDARY OUTCOMES:
Change in AHI | up to 5 hours
  Change in AHI in the "ON" versus "OFF" period
Percentage difference of time (minutes) per hour of sleep with loud snoring | up to 5 hours
  Percentage difference of time (minutes) per hour of sleep with loud snoring (≥40) in the "ON" versus "OFF" phase
Change in the number of arousals and awakenings in the "ON" versus "OFF" phase | up to 5 hours
  Change in the number of arousals and awakenings in the "ON" versus "OFF" phase
Difference in the mean oxygen saturation levels | up to 5 hours
  Difference in the mean oxygen saturation levels in the "ON" versus "OFF" phase
Number of patients with successful snoring reduction | up to 5 hours
  ≥ 25% reduction in snoring intensity in the "OFF" versus the "ON" period.

OTHER OUTCOMES:
Incidence of adverse events, serious adverse events, device deficiencies and unanticipated adverse device effects | up to 96 hours
  Safety and tolerability of intervention
Percent of the time the ZENS Device was adhered to the participant | up to 12 hours
  % time worn during entire study (awake and asleep)
Tolerability of the ZENS Device | up to 12 hours
  % of time worn during sleep

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Povitz, MD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - University of Calgary, FMC Sleep Centre, Calgary, Alberta
  - Tranq Sleep Centre, Cranbrook, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Zennea Technologies website — http://www.zenneatech.com/